CLINICAL TRIAL: NCT07036549
Title: Impact of Preoperative Sleep Quality and Anxiety on Postoperative Outcomes in Abdominal Gynecologic Cancer Surgery: A Prospective Observational Study
Brief Title: Impact of Preoperative Sleep Quality and Anxiety on Postoperative Outcomes in Abdominal Gynecologic Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Izmir City Hospital (Other Government)
Responsible Party: Principal Investigator, Celal Akdemir, MD, Izmir City Hospital
Other Study IDs: ISHSLANXPAIN
Record Dates: First submitted 2025-06-17; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-02

CONDITIONS: Gynecologic Neoplasms
Keywords: Sleep Quality; Anxiety; Postoperative Pain; Gynecologic Cancer Surgery; Preoperative Assessment; Patient Outcomes; Psychological Stress; Hospital Stay
MeSH Terms: conditions — Genital Neoplasms, Female; Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Pain, Postoperative; Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Patients undergoing abdominal gynecologic cancer surgery were prospectively observed for postoperative outcomes including pain, complications, analgesic requirement, and hospital stay. Preoperative sleep quality and anxiety levels were measured and analyzed in relation to clinical outcomes.

SUMMARY:
This prospective observational study aims to evaluate the effects of preoperative sleep quality and anxiety levels on postoperative outcomes in patients undergoing abdominal gynecologic cancer surgery. A total of 72 patients were included and assessed using the Pittsburgh Sleep Quality Index (PSQI) and the Beck Anxiety Inventory (BAI) prior to surgery. Postoperative outcomes including pain scores (measured by the Numeric Rating Scale), complication rates, additional analgesic use, and length of hospital stay were recorded. The findings suggest that poor sleep quality and high anxiety levels prior to surgery are significantly associated with higher postoperative pain, increased complication rates, and prolonged hospital stay. These results emphasize the importance of preoperative psychological evaluation and supportive interventions to improve perioperative care in gynecologic oncology.

DETAILED DESCRIPTION:
This prospective observational study was conducted between February and May 2025 at a tertiary gynecologic oncology center. The aim was to evaluate the association between preoperative sleep quality and anxiety levels with postoperative outcomes in patients undergoing open abdominal surgery for gynecologic cancer.

Eligible participants were women aged 18 years or older who were scheduled for elective laparotomy with general anesthesia. Patients with psychiatric disorders, major neurological conditions, or incomplete postoperative data were excluded.

Sleep quality was assessed preoperatively using the Pittsburgh Sleep Quality Index (PSQI), and anxiety was measured using the Beck Anxiety Inventory (BAI). Patients with a PSQI score ≥5 were classified as having poor sleep quality, and those with BAI scores ≥16 were classified as having high anxiety.

Postoperative pain was evaluated using the Numeric Rating Scale (NRS) at 0, 4, 8, 12, and 24 hours after surgery. Additional analgesic requirements, early postoperative complications (e.g., surgical site infection, ileus, nausea-vomiting, atelectasis), and length of hospital stay were recorded.

The study also examined potential psychosocial contributors such as mobile phone use during sleep, internet-based health information seeking, and patients' satisfaction with preoperative counseling using a structured Likert scale.

All data were collected via face-to-face interviews and hospital records. Statistical analyses included Mann-Whitney U test, chi-square test, and Spearman correlation coefficients. The study was approved by the Institutional Ethics Committee (Approval No: 2025/38), and all participants provided written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥18 years
* Diagnosed with gynecologic malignancy
* Scheduled for elective abdominal surgery (laparotomy)
* Able to provide informed consent
* Completed preoperative sleep and anxiety assessments

Exclusion Criteria:

* History of psychiatric or cognitive disorders interfering with questionnaire participation
* Emergency surgical procedures
* Incomplete follow-up data within 30 days postoperatively
* Patients admitted for inpatient observation prior to surgery
* Major previous pelvic surgery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only biologically female individuals undergoing gynecologic cancer surgery were eligible to participate.
Study Population: Female patients aged 18 years or older undergoing abdominal surgery for gynecologic malignancies at a tertiary oncology center between February and May 2025.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Score (Numeric Rating Scale) | Postoperative Day 1 (within 24 hours after surgery)
  Postoperative pain will be assessed using the Numeric Rating Scale (NRS) at 0, 4, 8, 12, and 24 hours after surgery. Higher scores indicate greater pain intensity.

SECONDARY OUTCOMES:
Postoperative Complication Rate | Up to 30 days after surgery
  Incidence of postoperative complications including surgical site infection, ileus, nausea-vomiting, and atelectasis recorded within 30 days after surgery.
Additional Analgesic Requirement | Postoperative Day 1 (within 24 hours after surgery)
  Requirement for rescue analgesics (non-protocol) within the first 24 hours postoperatively.
Length of Hospital Stay | From day of surgery until discharge (mean: 4.2 days)
  Duration of postoperative hospitalization measured in days from the day of surgery until the day of discharge, based on electronic medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Celal Akdemir, md, Principal Investigator — Izmir City Hospital
Locations (1):
- İzmir City Hospital, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akdemir C, Turan SA, Balci MF, Ozen S, Seker N, Bayramoglu D, Bayramoglu Z, Sanci M. Preoperative sleep quality and anxiety as predictors of postoperative pain and recovery in Gynecologic oncology surgery: A prospective observational study. J Psychosom Res. 2026 Feb;201:112496. doi: 10.1016/j.jpsychores.2025.112496. Epub 2025 Dec 11. PMID 41389754